CLINICAL TRIAL: NCT00951535
Title: A Prospective Phase II Dose Escalation Study Using IMRT for High Risk N0M0 Prostate Cancer
Brief Title: A Prospective Phase II Dose Escalation Study Using IMRT for High Risk N0 M0 Prostate Cancer. ICORG 08-17
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-17 ICORG; CTRIAL-IE 08-17 (Other: Cancer Trials Ireland)
Record Dates: First submitted 2009-08-01; First posted 2009-08-04 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Image-Guided; Radiotherapy, Intensity-Modulated

ARMS (1):
- Arm A (Other): Treatment will be delivered in 1.8 Gy fractions; dose escalation will be in 1.8 Gy increments from 75.6 Gy to a maximum 81 Gy.
  Interventions: Other: questionnaire administration; Procedure: quality-of-life assessment; Radiation: image-guided radiation therapy; Radiation: intensity-modulated radiation therapy; Radiation: radiation therapy treatment planning/simulation

INTERVENTIONS:
Other: questionnaire administration
Procedure: quality-of-life assessment
Radiation: image-guided radiation therapy
Radiation: intensity-modulated radiation therapy
Radiation: radiation therapy treatment planning/simulation

SUMMARY:
This is a prospective, phase II non-randomised controlled clinical study. Dose escalation will be implemented using 1.8 Gy increments from baseline 75.6 Gy. Patients' RT prescription may be escalated up to max 81 Gy once dose volume constraints are adhered to.

All patients will be treated using the participating institution's standard rectal preparation protocol, bladder-filling protocol and appropriate immobilisation device(s).

Cone beam CT on-treatment imaging is recommended for this study. However, the use of individual institutional imaging equipment and techniques is permitted.

Acute GU/GI toxicities will be assessed weekly during treatment.

GU/GI toxicities will also be assessed 2 months post RT, 8 months post RT and 6 monthly thereafter to year nine and in line with the participating institution's standard routine follow-up (FU) thereafter.

Translational sub-studies (optional), only apply to patients who are consented prior to commencement of hormone therapy at centres participating in the translational sub-study. Patients at centres participating in the translational sub-studies will be given the option of participating in sub-study 1 (Proteomic Analysis), sub-study 2 (Raman spectroscopic analysis), or both (sample collection will not be mandatory).

DETAILED DESCRIPTION:
Primary Objective:

To determine if dose escalated IMRT for high risk localised prostate cancer can provide PSA relapse free survival similar to that reported by Memorial Sloan Kettering (Alicikus et al 2011).

Sub-Study 1 (Proteomic Analysis):

To use proteomic analysis of sequential blood and urine samples to detect changes in profiles that may predict outcome and identify prognostic biochemical markers of early disease progression and/ or toxicity. The unique molecular signatures may also allow the identification of targets for therapeutic intervention.

To undertake, where possible, other biochemical analyses including mRNA, miRNA and metabolite profiling.

Sub-Study 2 (Raman spectroscopic analysis):

To investigate a new approach to prediction of radiation response, based on biochemical fingerprinting

Secondary Objectives:

* Overall survival and disease-free survival rates.
* To evaluate the significance of published prognostic/ stratification factors such as the UCSF-CAPRA score and assess their application to the data from this study.
* To achieve the maximum dose escalation (up to 81Gy). This will be assessed as the percentage of patients that receive each dose level for all categories (dose increments of 1.8 Gy from 75.6 Gy up to max 81 Gy).
* The incidence and severity of acute and late GU, GI and erectile dysfunction toxicities will be described, and correlated with DVH parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing a radical course of RT for high-risk disease (defined according to the National Comprehensive Cancer Network Practice Guidelines in Oncology v.1 as one or more of the NCCN high risk criteria > or equal to T3, > or equal to Gleason 8, PSA > 20ng/ml)
2. Only patients requiring neo-adjuvant / adjuvant hormonal therapy will be included in this study
3. Absence of distant metastases as demonstrated by history and physical examination, FBC, screening profile including liver function tests, PSA and bone scan
4. All patients must have an MRI/CT of the prostate and pelvis to investigate the nodal status and precise T-stage. This MRI/CT scan must be performed prior to commencement of hormonal therapy. Suspicious nodes need to be histologically proven to be benign before the patient can be included in the study). M0 on staging.
5. No previous surgery for urinary conditions except TURP or TRUS
6. KPS > or equal to 60
7. Age >18 years
8. Provision of written informed consent in line with ICH-GCP guidelines

Exclusion Criteria:

1. Previous RT to the pelvic region
2. The patient has nodal involvement or it is decided to electively treat pelvic lymph nodes
3. The patient has had a bilateral orchidectomy
4. The patient has previously received a full course of hormonal treatment for his prostate cancer
5. The patient has or has had other malignancies within the last 5 years (non-melanoma skin cancer is permitted)
6. Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the trial or if it is felt by the research/ medical team that the patient may not be able to comply with the protocol
7. Patients who have had a prostatectomy
8. The presence of hip prostheses

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2009-07-20 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Biochemical Failure Free survival | 7-9 years median follow-up

SECONDARY OUTCOMES:
Overall survival and disease free survival rates | 5-7 years follow-up
Maximum dose escalation | 9 years follow-up
The incidence and severity of Genito-urinary (GU), Gastro-intestinal (GI) and erectile dysfunction (ED) toxicities (graded by NCI CTCAE Version 3.0) will be analysed and correlated with dose volume histogram (DVH) parameters. | 9 years follow-up

OTHER OUTCOMES:
Identify prognostic and biochemical markers of early disease progression (Sub-Study 1) | 9 years follow-up
  To detect changes in profiles that may predict outcome and identify prognostic and biochemical markers of early disease progression in accordance with the primary and secondary objectives using Proteomic Analysis of sequential blood and urine samples.
Develop a platform for endpoint prediction using Raman spectroscopy and machine learning (Sub-Study 2) | 9 years follow-up
  Raman spectra will be recorded from both lymphocytes and sera to produce a library of spectral measurements in patients pre- and post-treatment. Established methodologies for the assessment of the patient radiosensitivity (G2 assay, DNA damage assays and gene expression profiling), will be used in parallel with advanced multivariate and machine learning methodologies to develop a platform for prediction of such endpoints using Raman spectra of the cellular and plasma fraction of the patient blood.

CONTACTS AND LOCATIONS:
Overall Officials: John Gerard Armstrong, MD, MB, MRCPI, Principal Investigator — SLRON St Luke's Hospital
Locations (5):
- Ireland (5):
  - Cork University Hospital, Cork
  - SLRON St Luke's Hospital, Dublin
  - Beacon Hospital, Dublin
  - SLRON St James's Hospital, Dublin
  - SLRON, Beaumont Hospital, Dublin

REFERENCES:
- [Background] Medipally DK, Maguire A, Bryant J, Armstrong J, Dunne M, Finn M, Lyng FM, Meade AD. Development of a high throughput (HT) Raman spectroscopy method for rapid screening of liquid blood plasma from prostate cancer patients. Analyst. 2017 Apr 10;142(8):1216-1226. doi: 10.1039/c6an02100j. PMID 28001146
- [Background] Medipally DKR, Nguyen TNQ, Bryant J, Untereiner V, Sockalingum GD, Cullen D, Noone E, Bradshaw S, Finn M, Dunne M, Shannon AM, Armstrong J, Lyng FM, Meade AD. Monitoring Radiotherapeutic Response in Prostate Cancer Patients Using High Throughput FTIR Spectroscopy of Liquid Biopsies. Cancers (Basel). 2019 Jul 2;11(7):925. doi: 10.3390/cancers11070925. PMID 31269684
- [Background] Cagney DN, Dunne M, O'Shea C, Finn M, Noone E, Sheehan M, McDonagh L, O'Sullivan L, Thirion P, Armstrong J. Heterogeneity in high-risk prostate cancer treated with high-dose radiation therapy and androgen deprivation therapy. BMC Urol. 2017 Aug 1;17(1):60. doi: 10.1186/s12894-017-0250-2. PMID 28764689
- [Derived] Meade AD, Maguire A, Bryant J, Cullen D, Medipally D, White L, McClean B, Shields L, Armstrong J, Dunne M, Noone E, Bradshaw S, Finn M, Shannon AM, Howe O, Lyng FM. Prediction of DNA damage and G2 chromosomal radio-sensitivity ex vivo in peripheral blood mononuclear cells with label-free Raman micro-spectroscopy. Int J Radiat Biol. 2019 Jan;95(1):44-53. doi: 10.1080/09553002.2018.1451006. Epub 2018 Mar 29. PMID 29528761